CLINICAL TRIAL: NCT06762691
Title: Cranial Remolding Orthosis Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Otto Bock HealthCare LP (Industry)
Responsible Party: Sponsor
Other Study IDs: OB114
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Plagiocephaly; Brachycephaly; Asymmetric Head
Keywords: CRO; MyCRO; Cranial Helmet; Cranial Orthosis; Cranial Remolding Orthosis
MeSH Terms: conditions — Plagiocephaly; Craniosynostoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Plagiocephaly: Infants diagnosed with plagiocephaly who have been scanned for a cranial remolding orthosis
  Interventions: Device: MyCRO Band; Device: Traditional CRO
- Brachycephaly: Infants diagnosed with brachycephaly who have been scanned for a cranial remolding orthosis
  Interventions: Device: MyCRO Band; Device: Traditional CRO

INTERVENTIONS:
Device: MyCRO Band — A 3D-printed cranial remolding orthosis
Device: Traditional CRO — A traditionally manufactured cranial remolding orthosis such as the Orthomerica Starband

SUMMARY:
A registry of infants fitted with a cranial remolding orthosis.

DETAILED DESCRIPTION:
The intention of the CRO registry is to gather real-world data of traditional and 3D-printed cranial remolding orthoses to compare outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been evaluated and successfully scanned for a MyCRO Band or similar CRO
* Patient's parent(s) or legal guardian(s) are able to communicate, provide feedback, understand and follow instructions during the course of the registry.
* Parent(s) or legal guardian(s) are willing to provide informed consent.

Exclusion Criteria:

* Patient is geographically inaccessible to comply and participate in the registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants who have been scanned and fitted with a cranial remolding orthosis
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Asymmetry Index | Baseline to final follow up visit (est. 6 months)
  Correction in Cranial Vault Asymmetry Index (Plagiocephaly) or Cephalic Index (Brachycephaly)

SECONDARY OUTCOMES:
Orthosis Utilization | Baseline to final follow up visit (est. 6 months)
  Orthosis wear time will be measured from an embedded sensor
QUEST 2.0 | Final follow up visit (est. 6 months)
  Quebec User Evaluation of Satisfaction with Assistive Technology 2.0

OTHER OUTCOMES:
Cranial Temperature | Baseline to final follow up visit (est. 6 months)
  Average temperature of the infant's head will be assessed by an embedded temperature sensor
Impact of delays on correction of asymmetry | Baseline to final follow up visit (est. 6 months)
  Percent reduction of asymmetry correction when delivery is delayed more than two weeks
Duration of therapy | Baseline to final follow up visit (est. 6 months)
  Average amount of time, in months, that the CRO was used
Impact of torticollis on compliance | Baseline to final follow up visit (est. 6 months)
  Percent reduction of wear time when torticollis is severe
Frequency of additional fittings | Baseline to final follow up visit (est. 6 months)
  Measuring the number of times the orthosis had to be refitted to accommodate changes in head shape

CONTACTS AND LOCATIONS:
Locations (1):
- Wright & Filippis, Madison Heights, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plans have been made to share IPD